CLINICAL TRIAL: NCT02486757
Title: Investigation of Female Reproductive Hormone Dynamics During Adolescence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013P-000513
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-06

CONDITIONS: Menstruation Disturbances
MeSH Terms: conditions — Menstruation Disturbances | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Experimental): estradiol 50 mcg transdermal patch x 7 days oral micronized progesterone 0.5 mg/kg/dose TID x 7 days
  Interventions: Drug: micronized progesterone; Drug: transdermal estradiol

INTERVENTIONS:
Drug: micronized progesterone
Drug: transdermal estradiol

SUMMARY:
Irregular menstrual cycles are common in girls for several years after their first menstrual period. The cause of abnormal menstrual cycles during this time is not well-understood. The purpose of this study is to: 1) monitor girls during a menstrual cycle (with blood and urine sampling and serial pelvic ultrasounds) to identify those girls who do not ovulate (release of an egg from the ovary), and 2) determine whether cycles can be corrected by treating girls with a short course of low-dose estrogen and progesterone.

ELIGIBILITY:
Inclusion Criteria:

* no more than 3 ½ years postmenarchal

Exclusion Criteria:

* Subjects currently on or previously treated with medications that may affect reproductive hormones (eg birth control pills).
* Subjects with severe acne or hirsutism
* Subjects who exercise excessively (running > 20 miles/week or its equivalent)
* Subjects with any of the following medical conditions: diabetes, hypertension, hyperlipidemia, valvular heart disease, lupus, rheumatoid arthritis, migraine headaches with aura, undiagnosed breast mass, inflammatory bowel disease, gallbladder disease, sickle cell disease, or thrombophilia.
* Current smoker
* History of deep venous thrombosis or pulmonary embolism in subject or first-degree relative

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Hall, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Reproductive Endocrine Unit, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortega MT, Carlson L, McGrath JA, Kangarloo T, Adams JM, Sluss PM, Lambert-Messerlian G, Shaw ND. AMH is Higher Across the Menstrual Cycle in Early Postmenarchal Girls than in Ovulatory Women. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1762-71. doi: 10.1210/clinem/dgaa059. PMID 32016427
- [Derived] Sun BZ, Kangarloo T, Adams JM, Sluss P, Chandler DW, Zava DT, McGrath JA, Umbach DM, Shaw ND. The Relationship Between Progesterone, Sleep, and LH and FSH Secretory Dynamics in Early Postmenarchal Girls. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2184-2194. doi: 10.1210/jc.2018-02400. PMID 30649404
- [Derived] Sun BZ, Kangarloo T, Adams JM, Sluss PM, Welt CK, Chandler DW, Zava DT, McGrath JA, Umbach DM, Hall JE, Shaw ND. Healthy Post-Menarchal Adolescent Girls Demonstrate Multi-Level Reproductive Axis Immaturity. J Clin Endocrinol Metab. 2019 Feb 1;104(2):613-623. doi: 10.1210/jc.2018-00595. PMID 30289507

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional: estradiol 50 mcg transdermal patch x 7 days oral micronized progesterone 0.5 mg/kg/dose TID x 7 days
  micronized progesterone
  transdermal estradiol
Period: Overall Study
Arm/Group | Interventional
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interventional
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Ovulation in Cycle 2
Description: serum progesterone > 3 ng/ml or presence of corpus luteum on pelvic ultrasound
Time Frame: 20-40 days
Population: subjects with sufficient data in cycle to determine ovulatory/anovulatory status
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 5
Participants
  ovulatory | 3
  anovulatory | 2

ADVERSE EVENTS:
Arm/Group | Interventional
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No